CLINICAL TRIAL: NCT04378452
Title: Assessment of the Psycho-social Impact of COVID-19 Outbreak (COM-COVID)
Brief Title: Assessment of the Psycho-social Impact of COVID-19 Outbreak
Acronym: COM-COVID
Status: Completed | Type: Observational
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Anaxomics SL (Unknown); Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other); Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Other Study IDs: COM-COVID
Record Dates: First submitted 2020-04-15; First posted 2020-05-07 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV 2; COVID-19; Quality of Life; Mental Health Wellness 1; Social Distance; SARS (Disease); Psychological
Keywords: SARS-CoV-2; COVID-19; psycho-social impact; mental health; infectious diseases
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Disease; Psychological Well-Being; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COM-COVID cohort: Individuals of >16 years old evaluated during the COVID-19 outbreak by an anonymous survey and willing to respond. Expected timeframe for the collection of completed surveys: March 31th, 2020-September 30th, 2020]
  Interventions: Behavioral: COM-COVID anonimous survey

INTERVENTIONS:
Behavioral: COM-COVID anonimous survey — Anonimous e-survey administered to the general population by sharing it through social and mass media, including questions on sociodemographic data, physical symptoms in the past 14 days compatible with SARS-CoV-2 infection, socio-economic impact of the COVID-19 outbreak and psychological impact of the COVID-19 outbreak and mental health status.

SUMMARY:
It has been shown in previous important outbreaks of infectious diseases that they have a huge impact on individuals and communities. The psychological effects of the illness itself and the traumatic experiences of loved ones are experienced by individuals and complete health systems. Added to this, the social ecosystem and family finances are also severely affected. After several months of the outbreak start and several weeks of quarantine and self-isolation, the emotional burden on the community has increased. Added to this, many of the confirmed cases are healthcare workers. In addition to the risk of infection, these front-line staff are exposed to high levels of stress and anxiety. This gets worse as the pressure on the health system increases, forcing them to deal with significant ethical issues.

To respond to all these issues, the research group led by Dr. Cris Vilaplana at the Germans Trias i Pujol Research Institute (IGTP), have launched a questionnaire to ask the public, including health professionals, how are they being affected by the pandemic, not only in relation to their health but in terms of their emotional wellbeing and their family finances. The project is an initiative of the SMA-TB consortium (IGTP and Anaxomics) to fight against COVID-19. The Fundació Lluita contra la SIDA is also collaborating in the project. The survey is based on questions related to depression, anxiety, stress, and post-traumatic stress disorder, which have already been used in other epidemic outbreaks and in disaster situations, but it also includes questions adapted to the current situation.

The survey (now available in 4 languages) has been designed to be shared using a snowball strategy, making possible for everybody to participate and collaborate. The results obtained will initially help us to better understand the impact of the outbreak of COVID-19 on the general wellbeing of the population and health workers so that we can go on to develop strategies in coordination those in charge of administrations in order to adapt policies to people's real needs. The results of the study will be published in a scientific article and will be publicly available.

DETAILED DESCRIPTION:
In March 30, 2020, 78797 confirmed cases of SARS-CoV-2, 6528 deaths and 14709 recovered were reported in Spain[1]; 16157 cases and 1410 deaths recorded in Catalonia[2]. Case fatality (8%) is calculated on the registered cases, even if the actual mortality rate is uncertain as the total number of cases (including those undiagnosed and with mild symptoms) is unknown [3]. It is already a fact that there is local transmission of SARS-CoV-2 in the community. Everyone with a compatible respiratory condition is considered likely to be a case of SARS-CoV-2[4], despite that the etiological diagnosis cannot be made in this context of health emergency for all cases suspected, because of the lack of kits, personnel and saturation of the health system.

Other major outbreaks of infectious diseases as Ebola have demonstrated that there is an important impact on the individuals and the communities. Psychological effects of the disease itself as well as the traumatic experience on the beloved ones are seen at individual level. At community level, health services, social system and economic productivity are severely affected[5].

After 2 months weeks of first case reported in Spain and 2,5 weeks of the quarantine and self-isolation of the region of Catalonia, the emotional burden of the general community has increased. In previous studies in other countries in which the SARS-CoV-2 epidemics have precede ours, a non despicable impact on mental health and emotional burden has been reported as well as has been demonstrated in mass quarantines which have been implemented in other epidemics context [6-8]. Moreover, a certain level of anxiety has been reported as necessary to adopt recommended precautionary measures against infection outbreaks[9], and therefore to successfully implement public health interventions understanding the attitudes and measuring psychological impact on people should be mandatory.

On the other hand, in our setting by last report at 30th March 2020, 2600 of the confirmed cases in Catalonia are healthcare workers, representing the 16%. Besides their obvious increased risk of being infected, the healthcare workers facing the SARS-CoV-2 epidemics at frontline (emergency rooms, ICUs and other dept.) are put under a lot of stress and levels of anxiety. This is worse as the tension to the Health Systems increase, they needing to face important ethical dilemmas including triage of patients. Moreover, SARS epidemic proved not only that frontline healthcare workers suffered from chronic stress, but that this lasted at least for one year after the epidemics wave was over [10].

The aim of the present study is to assess the psychological and socio-economic impact of the COVID-19 epidemics, and we intend to do this on both the general population and the healthcare workers.

An anonymous online survey is been shared through social media networks (including telegram, whatsapp, twitter) in order to get as many responses as possible from individuals of >16 years old. For the healthcare workers subpopulation the questionnaire will be also be distributed via email, posters, institutional websites and other means deemed appropriate (in hospital or other healthcare settings). The anonymous online survey will include questions on sociodemographic data, physical symptoms in the past 14 days, socio-economic impact of the COVID-19 outbreak, psychological impact of the COVID-19 outbreak and mental health status (through questions related to depression, anxiety, stress and PSTD, which have been used in other studies). We will share the survey through social media using the snowball sampling. We will continuously share the survey in order to collect responses 6 months after the outbreak, to learn how much the impact of it can last.

The results obtained will allow us to:

* Understand more accurately the impact of the COVID-19 outbreak on general population wellbeing.
* Measuring the impact on the health-care workers subpopulation which is critical to cope outbreaks is important to design interventions for stress management and enchance infection-control measures and patient care.

The COM-COVID project is led by Dr. Cris Vilaplana (Institute for Health Science Research Germans Trias i Pujol (IGTP)). Dr. Vilaplana's team, mainly dedicated to the study of tuberculosis (https://unitatdetuberculosiexperimental.wordpress.com/), has been following a research line for the last 4 years measuring the quality of life of people in the context of infectious diseases so that they can study people suffering from them in a more holistic and humanistic way[11,12]. The project is an initiative of the SMA-TB consortium (https://www.smatb.eu/) (IGTP and Anaxomics) to fight against COVID-19. The Fundació Lluita contra la SIDA (https://www.flsida.org/en) is also collaborating in the project.

ELIGIBILITY:
Inclusion Criteria:

* age = or >16 years old
* accepting to participate in the project and filling in the survey questionnaire

Exclusion Criteria:

* age <16 years old
* non accepting to participate in the project and filling in the survey questionnaire

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The respondents to the survey can choose one of the following responses to the question: "Which gender do you identify with?": male, female, non binary, I prefer not to say
Study Population: All people >16 years old willing to participate in the COM-COVID survey study during the COVID-19 outbreak (period March 2020-September 2020).
Sampling Method: Non-Probability Sample
Enrollment: 56656 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Psychological impact of the outbreak, total score | Through study completion, an average of 1 year.
  Psychological impact of the outbreak, total score will be measured by the sum of the depression questions score, the anxiety questions score, the stress questions score and the PSTD questions score. The results will be given according to being part of general population and according to being part of the healthcare workers subpopulation. Responses will also be reported minimum per gender, age, country and postal code.Results will be represented by week of survey completion, and reported related to relevant dates (weeks of confinement, major announcements to the whole population by their Governments, etc.)
Psychological impact of the outbreak: depression questions score | Through study completion, an average of 1 year.
  The score will be calculated as the result of the sum of the points received per question, each question can be answered in a range of 1-4. The results will be given according to being part of general population and according to being part of the healthcare workers subpopulation. Responses will also be reported minimum per gender, age, country and postal code.Results will be represented by week of survey completion, and reported related to relevant dates (weeks of confinement, major announcements to the whole population by their Governments, etc.)
Psychological impact of the outbreak: anxiety questions score | Through study completion, an average of 1 year.
  The score will be calculated as the result of the sum of the points received per question, each question can be answered in a range of 1-4. The results will be given according to being part of general population and according to being part of the healthcare workers subpopulation. Responses will also be reported minimum per gender, age, country and postal code.Results will be represented by week of survey completion, and reported related to relevant dates (weeks of confinement, major announcements to the whole population by their Governments, etc.)
Psychological impact of the outbreak: stress questions score | Through study completion, an average of 1 year.
  The score will be calculated as the result of the sum of the points received per question, each question can be answered in a range of 1-4. The results will be given according to being part of general population and according to being part of the healthcare workers subpopulation. Responses will also be reported minimum per gender, age, country and postal code.Results will be represented by week of survey completion, and reported related to relevant dates (weeks of confinement, major announcements to the whole population by their Governments, etc.)
Psychological impact of the outbreak: PSTD questions score | Through study completion, an average of 1 year.
  The score will be calculated as the result of the sum of the points received per question, each question can be answered in a range of 0-4. The results will be given according to being part of general population and according to being part of the healthcare workers subpopulation. Responses will also be reported minimum per gender, age, country and postal code.Results will be represented by week of survey completion, and reported related to relevant dates (weeks of confinement, major announcements to the whole population by their Governments, etc.)
Descriptive statistics for the non-psychological questions | Through study completion, an average of 1 year.
  Percentages of response will be calculated according to the number of respondents per each response out of the total number of responses of each question. All results will be given according to the respondents being part of the whole cohort of respondents, according to being part of general population and according to being part of the healthcare workers subpopulation. Responses will also be reported per gender, age, country and postal code.

CONTACTS AND LOCATIONS:
Overall Officials: Cris Vilaplana, MD, PhD, Principal Investigator — Fundació Institut Germans Trias i Pujol
Locations (4):
- Spain (4):
  - Fundació Institut Germans Trias i Pujol, Badalona, Catalonia
  - Fundació Lluita contra la Sida (FLS, Fight AIDS Foundation), Badalona, Catalonia
  - Anaxomics biotech, Barcelona
  - Fundació Privada per a la Recerca i la Docència Sant Joan de Déu, Esplugues de Llobregat

IPD SHARING:
Plan to Share IPD: Undecided
Results and database could be available upon request.

REFERENCES:
- [Result] Farres J, Ruiz JL, Mas JM, Arias L, Sarrias MR, Armengol C, Cardona PJ, Munoz-Moreno JA, Vilaplana M, Arranz B, Usall J, Serrano-Blanco A, Vilaplana C. Identification of the most vulnerable populations in the psychosocial sphere: a cross-sectional study conducted in Catalonia during the strict lockdown imposed against the COVID-19 pandemic. BMJ Open. 2021 Nov 26;11(11):e052140. doi: 10.1136/bmjopen-2021-052140. PMID 34836903
- See also: COM-COVID project website — https://comcovid.wixsite.com/com-covid?lang=en
- See also: COM-COVID results -complete dataset results generated — https://doi.org/10.5281/zenodo.4608501